CLINICAL TRIAL: NCT02426879
Title: Esophagectomy for Patients With Esophageal Cancer and Cervical Lymph Node Metastases Node Study
Brief Title: Esophagectomy for Patients With Esophageal Cancer and Cervical Lymph Node Metastases
Acronym: Node
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Richard van Hillegersberg, prof Dr, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL48231.041.14
Record Dates: First submitted 2015-01-30; First posted 2015-04-27 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Cancer; Squamous Cell Carcinoma; Adenocarcinoma; Malignancy
Keywords: three-field lymphadenectomy; cervical metastases; esophagectomy
MeSH Terms: conditions — Neoplasms; Carcinoma, Squamous Cell; Adenocarcinoma | interventions — Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- surgery (Other): esophagectomy with three-field lymphnode dissection
  Interventions: Procedure: esophagectomy with three-field lymphnode dissection

INTERVENTIONS:
Procedure: esophagectomy with three-field lymphnode dissection — robot assisted thoraco-laparoscopic esophagectomy with three-field lymphnode dissection

SUMMARY:
There is no world-wide consensus on the oncological benefit versus increased morbidity associated with three field lymphadenectomy in patients with esophageal cancer and cervical lymph node metastases. In Asian countries, esophagectomy is commonly combined with a three field lymphadenectomy, including resection of cervical, thoracic and abdominal lymph nodes. However, in Western countries patients with cervical lymph node metastases are generally precluded from curative treatment.

DETAILED DESCRIPTION:
Objective: To assess the safety and feasibility of curative esophagectomy combined with three field lymphadenectomy after chemo-radiation in Western patients with resectable thoracic esophageal carcinoma and cervical lymph node metastases. Secondary objective is to determine the effect on survival and recurrence.

Study design: Mono centre prospective phase II single-arm feasibility study. Study population: Western patients diagnosed with resectable (cT1-4a, N1-3) intra thoracic esophageal carcinoma with histological or cytological proven cervical lymph node metastases in level III and/ or IV.

Intervention: Transthoracic esophageal resection combined with three field lymphadenectomy after neoadjuvant chemo-radiation.

Main study parameters/ endpoints: Primary outcome is the percentage of overall surgical complications grade 3b and higher as stated by the Modified Clavien-Dindo classification. Secondary outcomes are mortality, operation related events and postoperative recovery, including quality of life, disease free survival, overall survival and if applicable the location of recurrent disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma or adenocarcinoma of the esophagus.
* Surgical resectable carcinoma (T1-4a, N1-3) (table 1)
* Histologically/ cytologically proven resectable cervical lymph node metastases level III and/ or IV
* Age ≥ 18
* European Clinical Oncology Group (ECOG) performance status 0,1 or 2
* Written informed consent

Exclusion Criteria:

* Distant metastases
* Esophageal carcinoma < 3 cm beneath UES
* Carcinoma of the gastro-esophageal junction (GEJ) with major tumor in the gastric cardia (Siewert III)
* Former radiotherapy or chemotherapy for esophageal carcinoma
* Former radiotherapy precluding radiotherapy according the CROSS protocol
* Inadequate pulmonary function disabling transthoracic resection
* >10% loss of weight in the last six months
* Previous neck dissection
* New York heart association class III/IV and no history of active angina. Patients with a history of significant ventricular arrhythmia requiring medication or congestive heart failure. History of 2nd or 3rd degree heart blocks

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Safety measured by the percentage of overall postoperative complications grade 3b and higher as stated by the modified Clavien-Dindo classification (MCDC) | 5 years
  Safety is measured by the percentage of overall postoperative complications grade 3b and higher as stated by the modified Clavien-Dindo classification (MCDC)

SECONDARY OUTCOMES:
mortality | 5 years
  in-hospital mortality and 30- and 60 day mortality (absolute numbers/ percentages)
survival | 5 years
  5 year overall- and disease free survival.
quality of life measured by questionnaires (EORTC-QLQ_C30 and EORTC-QLQ_Oes18) | 10 years
  QoL is measured by questionnaires (EORTC-QLQ_C30 and EORTC-QLQ_Oes18)
operation related events 1 | 5 years
  duration of surgery (minutes)
operation related events 2 | 5 years
  reason for prolongation of surgery if applicable
operation related events 3 | 5 years
  unexpected events/ complications
operation related events 4 | 5 years
  bloodloss (ml) reason for conversion if applicable.
operation related events 5 | 5 years
  reason for conversion if applicable.
postoperative recovery | 5 years
  duration of intubation (days), length of ICU/ MCU stay(days), length of hospital stay (days),

OTHER OUTCOMES:
pathology results 1 | 5 years
  pTNM stage
pathology results 2 | 5 years
  site of tumour
pathology results 3 | 5 years
  length of tumour
pathology results 4 | 5 years
  type of tumour
pathology results 5 | 5 years
  gradation of tumour
pathology results 6 | 5 years
  margins of resection (R0, R1, R2)
pathology results 7 | 5 years
  mandard score
pathology results 8 | 5 years
  lymphnode status
pathology results 9 | 5 years
  vaso-invasion
pathology results 10 | 5 years
  perineural growth

CONTACTS AND LOCATIONS:
Overall Officials: Richard V Hillegersberg, Prof Dr, Principal Investigator — UMCU
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] van der Horst S, Weijs TJ, Braunius WW, Mook S, Mohammed NH, Brosens L, van Rossum PSN, Weusten BLAM, Ruurda JP, van Hillegersberg R. Safety and Feasibility of Robot-Assisted Minimally Invasive Esophagectomy (RAMIE) with Three-Field Lymphadenectomy and Neoadjuvant Chemoradiotherapy in Patients with Resectable Esophageal Cancer and Cervical Lymph Node Metastasis. Ann Surg Oncol. 2023 May;30(5):2743-2752. doi: 10.1245/s10434-022-12996-x. Epub 2023 Jan 27. PMID 36707482